CLINICAL TRIAL: NCT04951752
Title: Effect of the Transmuscular Quadratus Lumborum Block on Duration of Stay in Recovery: a Single-centre, Retrospective, Observational Study Based on Five Selected Randomised Controlled Trials
Brief Title: Effect of the Transmuscular Quadratus Lumborum Block on Duration of Stay in Recovery
Acronym: TQL_PACU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SOPRE-001
Record Dates: First submitted 2021-04-14; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Hemicolectomy, Active treatment: 2x30mL 0.375% Ropivacaine administered by way of transmuscular quadratus lumborum block
  Interventions: Drug: Ropivacaine injection
- Hemicolectomy, Placebo treatment: 2x30mL isotonic saline administered by way of transmuscular quadratus lumborum block
- Nephrectomy, Active treatment: 2x30mL 0.375% Ropivacaine administered by way of transmuscular quadratus lumborum block
  Interventions: Drug: Ropivacaine injection
- Nephrectomy, Placebo treatment: 2x30mL isotonic saline administered by way of transmuscular quadratus lumborum block
- Percutaneous nephrolithotomy, Active treatment: 1x30mL 0.75% Ropivacaine administered by way of transmuscular quadratus lumborum block
  Interventions: Drug: Ropivacaine injection
- Percutaneous nephrolithotomy, Placebo treatment: 1x30mL isotonic saline administered by way of transmuscular quadratus lumborum block
- Hysterectomy, Active treatment: 2x30mL 0.375% Ropivacaine administered by way of transmuscular quadratus lumborum block
  Interventions: Drug: Ropivacaine injection
- Hysterectomy, Placebo treatment: 2x30mL isotonic saline administered by way of transmuscular quadratus lumborum block
- Elective Caesarean section, Active treatment: 2x30mL 0.375% Ropivacaine administered by way of transmuscular quadratus lumborum block
  Interventions: Drug: Ropivacaine injection
- Elective Caesarean section, Placebo treatment: 2x30mL isotonic saline administered by way of transmuscular quadratus lumborum block

INTERVENTIONS:
Drug: Ropivacaine injection — Transmuscular quadratus lumborum block - active
  Other Names: Transmuscular quadratus lumborum block
  Groups: Elective Caesarean section, Active treatment; Hemicolectomy, Active treatment; Hysterectomy, Active treatment; Nephrectomy, Active treatment; Percutaneous nephrolithotomy, Active treatment

SUMMARY:
The study will review data collected in 5 previously completed randomised controlled trials with a new primary outcome: to assess whether administration of the transmuscular quadratus lumborum block has an impact on the time an individual patient stays in the postanaesthesia care unit and how much opioid is consumed during this specified time.

ELIGIBILITY:
Inclusion Criteria:

- Elective Surgery

Exclusion Criteria:

* Inability to cooperate
* Allergy to local anaesthetics or opioids
* Inability to understand Danish
* Regular intake of opioids
* Local infection at site of injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery (hemicolectomy, nephrectomy, percutaneous nephrolithiotomy, hysterectomy of caesarean section).
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Duration of recovery | 0-300 minutes
  Minutes from arrival in PACU to completed recovery (arrival until ready for departure)

SECONDARY OUTCOMES:
Total time spent in recovery | 0-300 minutes
  Minutes from arrival in PACU to actual departure time (arrival until actual departure)
Duration of stay at PACU after completed recovery | 0-300 minutes
  Minutes from completed recovery to actual departure from PACU
Total opioid consumption in PACU | 0-300 minutes
  Total amount of opioid administered, converted to Oral Morphine Equivalents
Highest pain score in PACU | 0-300 minutes
  Highest reported Numeric Rating Scale of pain during stay in recovery

CONTACTS AND LOCATIONS:
Overall Officials: Jens Børglum Neimann, MD, PhD, Study Director — Associate Professor, Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request

REFERENCES:
- [Background] Dam M, Hansen C, Poulsen TD, Azawi NH, Laier GH, Wolmarans M, Chan V, Bendtsen TF, Borglum J. Transmuscular quadratus lumborum block reduces opioid consumption and prolongs time to first opioid demand after laparoscopic nephrectomy. Reg Anesth Pain Med. 2021 Jan;46(1):18-24. doi: 10.1136/rapm-2020-101745. Epub 2020 Oct 26. PMID 33106280
- [Background] Hansen CK, Dam M, Steingrimsdottir GE, Laier GH, Lebech M, Poulsen TD, Chan VWS, Wolmarans M, Bendtsen TF, Borglum J. Ultrasound-guided transmuscular quadratus lumborum block for elective cesarean section significantly reduces postoperative opioid consumption and prolongs time to first opioid request: a double-blind randomized trial. Reg Anesth Pain Med. 2019 Jul 14:rapm-2019-100540. doi: 10.1136/rapm-2019-100540. Online ahead of print. PMID 31308263
- [Result] Dam M, Hansen CK, Poulsen TD, Azawi NH, Wolmarans M, Chan V, Laier GH, Bendtsen TF, Borglum J. Transmuscular quadratus lumborum block for percutaneous nephrolithotomy reduces opioid consumption and speeds ambulation and discharge from hospital: a single centre randomised controlled trial. Br J Anaesth. 2019 Aug;123(2):e350-e358. doi: 10.1016/j.bja.2019.04.054. Epub 2019 May 30. PMID 31153628